CLINICAL TRIAL: NCT04130061
Title: Safety and Feasibility Human Amniotic Membrane to Decrease Post Operative Atrial Fibrillation After Coronary Artery Bypass Grafting
Brief Title: Human Amniotic Membrane to Decrease Post Operative Atrial Fibrillation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Vikas Sharma, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00113483
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Randomized (Experimental)
  Interventions: Biological: Human Amniotic Membrane
- Control (No Intervention)

INTERVENTIONS:
Biological: Human Amniotic Membrane — Epicardial application of human amniotic membrane during cardiac surgery
  Arms: Randomized

SUMMARY:
This study will evaluate the application of hAM at the time of cardiac surgery to decrease inflammation and the subsequent substrate to reduce incidence of post-operative atrial fibrillation. Patients will randomized 1:1 to receive either hAM application or standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary elective CABG at the University of Utah Hospital
* Ability to provided informed consent and follow-up with protocol procedures

Exclusion Criteria:

* Patients in AF at the time of surgery
* Prior history of sternotomy
* Prior history of pericarditis
* Currently on aggressive antiarrhythmic therapy (does not include beta blockers)
* Patients with an implantable cardiac device (pacemaker, ICD, CRT-D)
* Ejection fraction <45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Sharma, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in a University hospital (inpatient, outpatient clinics) from October 2019 through May 2021
Pre-assignment Details: One participant was enrolled and randomized to receive the intervention, but they ultimately did not have the membrane placed due to a miscommunication in the OR. This is the reason that 27 participants were enrolled but the total number for analysis was 26.
Groups:
- Randomized: Patients undergoing isolated CABG who randomized to receive amniotic membrane
- Control: Patients undergoing isolated CABG who randomized to receive standard of care
Period: Overall Study
Arm/Group | Randomized | Control
Started | 13 | 14
Completed | 12 | 14
Not Completed | 1 | 0
Not completed — OR team forgot to request membrane | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized: Patients undergoing isolated CABG surgery who are randomized to receive amniotic membrane
- Control: Patients undergoing isolated CABG surgery who are randomized to receive standard of care
- Total: Total of all reporting groups
Arm/Group | Randomized | Control | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 64.91 [54 to 76] | 65.78 [49 to 81] | 65.38 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The AM applied epicardially will be assessed for signs of hyperacute rejection i.e. membrane changing color; cardiac tamponade or constriction assessed by echocardiogram and transmission of infectious diseases. The incidence of adverse events (AEs) will be reported as percentages, with two-sided 95% confidence intervals. Statistical comparisons of AEs between the AM treatment and the control group will be made using a chi-square, or Fisher's exact test, as appropriate (based on the minimum expected cell frequencies).
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Post Op Atrial Fibrillation Between Patients Who Receive hAM and Controls
Description: The number of patients with Post Op Atrial Fibrillation will be compared between the treatment and control group using mobile telemetry. This comparison will be analyzed using chi-square or Fisher's exact test as appropriate.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized | Control
Number analyzed (Participants) | 13 | 14
Participants | 5 | 6

3. Primary Outcome: proBNP (Serum) Between Groups at Time of Surgery
Description: Comparison of serum levels of proBNP between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 13
pg/mL | 198 (263) | 347 (523)

4. Primary Outcome: C-reactive Protein (Serum) Between Groups at Time of Surgery
Description: Comparison of serum levels of CRP between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 0.34 (0.32) | 0.39 (0.87)

5. Primary Outcome: Interleukin-6 (Serum) Between Groups at Time of Surgery
Description: Comparison of serum measurement of IL-6 between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 13
pg/mL | 2.25 (0.86) | 2.23 (0.83)

6. Primary Outcome: Tumor Necrosis Factor - Alpha (TNFa; Serum) Between Groups at Time of Surgery
Description: Comparison of serum levels of TNFa between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 13
pg/mL | 2.45 (1.56) | 3.63 (3.04)

7. Primary Outcome: proBNP (Serum) Between Groups at 24 Hours Post-op
Description: Comparison of serum proBNP levels between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 1922.83 (1017.9) | 2239.42 (2384.3)

8. Primary Outcome: C-reactive Protein (Serum) Between Groups at 24-hours Post-op
Description: Comparison of serum measurements of CRP between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 14.94 (5.94) | 10.66 (4.58)

9. Primary Outcome: Interleukin-6 (Serum) Between Groups at 24-hours Post-op
Description: Comparison of IL-6 serum levels between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 26.95 (22.36) | 18.28 (12.03)

10. Primary Outcome: Tumor Necrosis Factor - Alpha (TNFa; Serum) Between Groups at 24 Hours Post-op
Description: Comparison of serum levels of TNFa between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 2.61 (1.22) | 2.87 (2.72)

11. Primary Outcome: proBNP (Serum) Between Groups at 48 Hours Post-op
Description: Comparison of serum levels of proBNP between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 6081.83 (5134.12) | 7750.35 (7474.25)

12. Primary Outcome: C-reactive Protein (Serum) Between Groups at 48 Hours Post-op
Description: Comparison of serum CRP levels between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 21.67 (8.18) | 15.71 (6.97)

13. Primary Outcome: Interleukin-6 (Serum) Between Groups at 48 Hours Post-op
Description: Comparison of IL-6 serum results between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 12.32 (10.01) | 14.39 (10.23)

14. Primary Outcome: Tumor Necrosis Factor - Alpha (Serum) Between Groups at 48 Hours Post-op
Description: Comparison of serum TNFa levels between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 2.34 (1.51) | 2.27 (1.09)

15. Primary Outcome: proBNP (Serum) Between Groups at 72 Hours Post-op
Description: Comparison of serum levels of proBNP between groups at 72 hour post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 2707.75 (925.9) | 449.71 (6191.8)

16. Primary Outcome: CRP (Serum) Between Groups at 72 Hours Post-op
Description: Comparison of serum levels of CRP between groups at 72 hour post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 9 | 11
mg/dL | 17.45 (5.95) | 14.21 (5.19)

17. Primary Outcome: Interleukin-6 (Serum) Between Groups at 72 Hours Post-op
Description: Comparison of IL-6 serum levels between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 9 | 11
pg/mL | 5.81 (4.15) | 10.38 (8.85)

18. Primary Outcome: TNFa (Serum) Between Groups at 72 Hours Post-op
Description: Comparison of TNFa serum levels between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 9 | 11
pg/mL | 2.12 (1.26) | 2.38 (1.56)

19. Primary Outcome: proBNP (Serum) Between Groups at Follow-up
Description: Comparison of serum levels of proBNP between groups at follow-up
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 10
pg/mL | 847 (505.79) | 1391.7 (1336.8)

20. Primary Outcome: CRP (Serum) Between Groups at Follow-Up
Description: Comparison of serum CRP levels between groups at follow-up
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 10
mg/dL | 0.975 (0.49) | 1.96 (3.61)

21. Primary Outcome: Interleukin-6 (Serum) Between Groups at Follow-up
Description: Comparison of IL-6 serum levels between groups at follow-up
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 10
pg/mL | 2.37 (1.06) | 6.86 (15.36)

22. Primary Outcome: TNFa (Serum) Between Groups at Follow-up
Description: Comparison of TNFa serum levels between groups at follow-up
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 10
pg/mL | 2.11 (1.16) | 3.11 (2.93)

23. Primary Outcome: proBNP (Pericardial Fluid) Between Groups at Time of Surgery
Description: Comparison of proBNP levels in pericardial fluid between groups at time of surgery (baseline)
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 13 | 14
pg/mL | 1039.6 (819.58) | 1771.07 (2332.54)

24. Primary Outcome: C-reactive Protein (Pericardial Fluid) Between Groups at Time of Surgery
Description: Comparison of CRP levels in pericardial fluid between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 0.34 (0.32) | 0.39 (0.87)

25. Primary Outcome: Interleukin-6 (Pericardial Fluid) Between Groups at Time of Surgery
Description: Comparison of IL-6 levels in pericardial fluid between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 11 | 13
pg/mL | 30.3 (26.17) | 59.9 (122.83)

26. Primary Outcome: Tumor Necrosis Factor - Alpha (Pericardial Fluid) Between Groups at Time of Surgery
Description: Comparison of TNFa in pericardial fluid between groups at the time of surgery (baseline).
Time Frame: Surgery
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 11 | 13
pg/mL | 2.81 (2.72) | 2.77 (2.46)

27. Primary Outcome: proBNP (Pericardial Fluid) Between Groups at 24 Hours Post-op
Description: Comparison of levels of proBNP in pericardial fluid between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 6081.83 (5134.12) | 7750.35 (7474.25)

28. Primary Outcome: C-reactive Protein (Pericardial Fluid) Between Groups at 24 Hours Post-op
Description: Comparison of CRP levels in pericardial fluid between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 4.54 (2.51) | 2.84 (2.05)

29. Primary Outcome: Interleukin-6 (Pericardial Fluid) Between Groups at 24 Hours Post-op
Description: Comparison of IL-6 levels in pericardial fluid between groups at 24 hours post-op
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 4 | 7
pg/mL | 88823.8 (51901.4) | 67217.8 (48407.4)

30. Primary Outcome: Tumor Necrosis Factor - Alpha (Pericardial Fluid) Between Groups at 24 Hours Post-op
Description: Comparison of TNFa in pericardial fluid between groups at 24 hours post-op.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 11 | 13
pg/mL | 8.58 (5.61) | 10.35 (8.04)

31. Primary Outcome: proBNP (Pericardial Fluid) Between Groups at 48 Hours Post-op
Description: Comparison of proBNP levels in pericardial fluid between groups at 48 hours post-op.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
pg/mL | 8823.4 (9286.9) | 10027.57 (7189.94)

32. Primary Outcome: C-reactive Protein (Pericardial Fluid) Between Groups at 48 Hours Post-op
Description: Comparison of CRP levels in pericardial fluid between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 14
mg/dL | 6.8 (3.72) | 4.9 (2.52)

33. Primary Outcome: Interleukin-6 (Pericardial Fluid) Between Groups at 48 Hours Post-op
Description: Comparison of IL-6 levels in pericardial fluid between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 5 | 9
pg/mL | 64370.14 (57497) | 45839.95 (43229.37)

34. Primary Outcome: Tumor Necrosis Factor - Alpha (Pericardial Fluid) Between Groups at 48 Hours Post-op
Description: Comparison of TNFa levels in pericardial fluid between groups at 48 hours post-op
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 12 | 13
pg/mL | 8.3 (7.81) | 8.03 (5.34)

35. Primary Outcome: proBNP (Pericardial Fluid) Between Groups at 72 Hours Post-op
Description: Comparison of proBNP levels in pericardial fluid between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 11
pg/mL | 3895.5 (1458.8) | 8423 (5911.3)

36. Primary Outcome: C-reactive Protein (Pericardial Fluid) Between Groups at 72 Hours Post-op
Description: Comparison of CRP levels in pericardial fluid between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 8 | 11
mg/dL | 8.53 (3.89) | 6.35 (3.1)

37. Primary Outcome: Interleukin-6 (Pericardial Fluid) Between Groups at 72 Hours Post-op
Description: Comparison of IL-6 levels in pericardial fluid between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 3 | 8
pg/mL | 9296.6 (9514) | 25316.6 (39863.65)

38. Primary Outcome: Tumor Necrosis Factor - Alpha (Pericardial Fluid) Between Groups at 72 Hours Post-op
Description: Comparison of TNFa levels in pericardial fluid between groups at 72 hours post-op
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized | Control
Number analyzed (Participants) | 7 | 10
pg/mL | 12.32 (13.44) | 8.38 (4.41)

ADVERSE EVENTS:
Time Frame: 30 days post-hospital discharge
Arm/Group | Randomized | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04130061/Prot_SAP_000.pdf